CLINICAL TRIAL: NCT04641637
Title: Substudy of Protocol TACE Emulsion Versus Suspension (NCT03268499): Interconnection of Arterial Tumor Feeders Through Tumor Sinusoid in Hepatocellular Carcinoma(HCC): In-vivo Proof of Concept and Clinical Implication
Brief Title: Substudy: Interconnection of Arterial Tumor Feeders Through Tumor Sinusoid in HCC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Simon Yu, Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VIR-20-12
Record Dates: First submitted 2020-11-18; First posted 2020-11-24 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Selective catheterization of segmental or more peripheral arteries in TACE (Other): From the digital subtraction angiography (DSA), the number of arterial tumor feeders to the HCC is identified. One or more feeder(s) is to be catheterized for delivery of therapeutic agent using a 2.4 French microcatheter (Merit Maestro, Merit Medical Systems, Utah, USA), and the other feeder(s) is occluded with a balloon catheter using 0.1 to 0.2mL diluted contrast for inflation (4mm x 10mm Temporary Occlusion Balloon Catheter, Occlusafe, Terumo Clinial Supply, Gifu, Japan). The occlusion target could be a feeder or a common trunk leading to a number of feeders.
  Interventions: Procedure: TACE

INTERVENTIONS:
Procedure: TACE — Through a 7 French sheath placed through a single femoral arterial puncture, a guide catheter (Cobra 1 Guide Catheter, Mach 1, Boston Scientific Corporation, Marlborough, USA) is placed at the coeliac axis. From the digital subtraction angiography (DSA), the number of arterial tumor feeders to the HCC is identified. One or more feeder(s) is to be catheterized for delivery of therapeutic agent using a 2.4 French microcatheter (Merit Maestro, Merit Medical Systems, Utah, USA), and the other feeder(s) is occluded with a balloon catheter using 0.1 to 0.2mL diluted contrast for inflation (4mm x 10mm Temporary Occlusion Balloon Catheter, Occlusafe, Terumo Clinial Supply, Gifu, Japan). The occlusion target could be a feeder or a common trunk leading to a number of feeders. The therapeutic agent was delivered under fluoroscopic control until the vasculature of the whole tumors is entirely filled, which was assessed with DSA and non-contrast CT performed at the completion of the procedure.

SUMMARY:
It is postulated that all arterial tumor feeders supplying a HCC tumor are interconnected with each other through the tumor sinusoid, such that when one of the feeders is catheterized for delivery of a liquid embolic agent, the whole tumor sinusoid will be embolized, if the arterial blood flow in all the other feeders are stopped temporarily to create a negative pressure gradient.

DETAILED DESCRIPTION:
Selective catheterization of segmental or more peripheral arteries in the procedure of transarterial treatment could be crucial in making a significant difference in survival outcome (1). Subsegmental chemoembolization (TACE) leading to portal vein visualization is associated with a higher chance of complete response (2), and complete response is a robust predictor of better overall survival (3). Selective TACE might also help to preserve liver function because TACE damages liver parenchyma and repeated TACE could lead to deterioration in liver function (4). In a procedure of ultra-selective TACE, each of the arterial tumor feeders is supposed to be catheterized for complete treatment of the whole tumor when there are multiple tumor feeders (5), it could be time consuming and technically challenging to achieve catheterize all the tumor feeders at a sub-subsegmental level when difficult arterial anatomy is encountered, even with the guidance of a automated tumor-feeders detection software (6). In the angioarchitecture of HCC, arterial tumor feeders lead to tumor sinusoid which is an interconnected network of vascular channel within the tumor substance (7). It is postulated that all arterial tumor feeders supplying a HCC tumor are interconnected with each other through the tumor sinusoid, such that when one of the feeders is catheterized for delivery of a liquid embolic agent, the whole tumor sinusoid will be embolized, if the arterial blood flow in all the other feeders are stopped temporarily to create a negative pressure gradient.

ELIGIBILITY:
Inclusion criteria Child-Pugh grade A, HCC diagnosed with typical arterial enhancement and portal washout patterns on contrast enhanced CT or MRI, solitary tumor, hypervascularity, well-defined margin, size ≤7cm, at least two arterial tumor feeders on CT scan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-06-30 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-04-28 (Actual)

PRIMARY OUTCOMES:
The completeness of coverage of the tumor vasculature by therapeutic agent at the completion of the treatment as evaluated on non-contrast CT scan | immediately after completion of procedure
  The completeness of coverage of the tumor vasculature by therapeutic agent at the completion of the treatment as evaluated on non-contrast CT scan

SECONDARY OUTCOMES:
Tumor response | 3 months
  Tumor response as evaluated on CT scan

CONTACTS AND LOCATIONS:
Overall Officials: Simon Yu, Professor, Principal Investigator — DIIR, CUHK, Hong Kong
Locations (1):
- Department of Imaging and Interventional Radiology, Prince of Wales Hospital, The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No